CLINICAL TRIAL: NCT01340066
Title: A Randomized, Double-blind, Parallel, Placebo-controlled Study for the Assessment of the Safety and Efficacy of UISH001 for the Symptomatic Improvement of Urinary Incontinence
Brief Title: Safety and Efficacy Study of a New Treatment for Symptoms of Urinary Incontinence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beech Tree Labs, Inc. (Industry)
Collaborators: Norwich Clinical Research Associates Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-2006-0081
Record Dates: First submitted 2011-04-18; First posted 2011-04-22 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; stress incontinence; urge incontinence; mixed incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UISH001 (Experimental)
  Interventions: Drug: UISH001
- Matching placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: UISH001 — sublingual dosing, 1 drop 3 times a day
  Arms: UISH001
Drug: matching placebo — sublingual dosing,1 drop 3 times a day
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to determine if a new drug treatment is effective for the treatment of symptoms of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women who have moderate to severe urge, stress or mixed Urinary Incontinence

Exclusion Criteria:

* Medical history of migraines, neurologic problems, swallowing disorder, stroke or severe depression.
* Medical history of heart failure, peripheral edema or moderate to severe asthma or chronic obstructive pulmonary disease (COPD)
* Certain restricted medications
* Any other condition that would interfere with the safety of the subject

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research, Rochester, New York
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three medical clinics during the study period of 05/06/2011 to 05/17/2012.
Pre-assignment Details: Participants entered a one week placebo run in period to fulfill inclusion/exclusion criteria before being randomized.
Groups:
- Placebo Run-In: All subjects entered a one week placebo run in period to qualify for the study.
- Placebo; UISH001: Subjects were randomized at Visit 2
Period: Placebo Run in Period
Arm/Group | Placebo Run-In | Placebo | UISH001
Started | 94 | 0 | 0
Completed | 67 (Completed run in period and were eligible for randomization) | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Screen Failures | 27 | 0 | 0
Period: 5 Week Double Blind Randomization Period
Arm/Group | Placebo Run-In | Placebo | UISH001
Started | 0 | 33 | 34
Completed | 0 | 28 | 31
Not Completed | 0 | 5 | 3
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics only for subjects that were randomized into the study.
Groups:
- Matching Placebo: At randomization at visit 2, subjects were treated with matching placebo.
- UISH001: At randomization at visit 2, subjects were treated with UISH001.
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | UISH001 | Total
Number analyzed (Participants) | 33 | 34 | 67
Age Continuous [Mean (Full Range); unit: Year]
  All subjects | 56.2 [36 to 92] | 52.6 [22 to 88] | 54.4 [22 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Decrease in Leakage Events of 30% or More.
Description: Incontinence events were recorded on a daily diary. Leaks were scored and tabulated for a daily score. These values were utilized to come up with total of leakage events during the double-blind treatment period.
Time Frame: Change from baseline after 4 weeks of treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: 1 drop Placebo sublingual 3 times/day
- UISH001: 1 drop UISH001 sublingual 3 times/day
Arm/Group | Placebo | UISH001
Number analyzed (Participants) | 33 | 34
Percentage of participants | 60.6 | 61.7
Statistical Analysis 1: Comparison: Placebo vs UISH001; Test type: Superiority or Other; p = .92, Chi-squared; Mean Difference (Final Values) = 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of informed consent to the end of the study (6 weeks)
Description: Subjects were queried concerning AEs at all visits.
Groups:
- Non-Randomized Subjects: Adverse Events (AEs) captured for subjects that were not randomized
- UISH001: Subjects were treated with UISH001 during double blind treatment period.
- Matching Placebo: Subjects were treated with matching placebo during double blind treatment period.
Arm/Group | Non-Randomized Subjects | UISH001 | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/27 | 15/34 | 7/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Randomized Subjects (N=27) | UISH001 (N=34) | Matching Placebo (N=33)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Randomized Subjects (N=27) | UISH001 (N=34) | Matching Placebo (N=33)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days